CLINICAL TRIAL: NCT06782932
Title: A Pilot Study Comparing Neoadjuvant and Adjuvant GVAX vs a Mutated KRAS Peptide Vaccine Given With Anti-PD-1 and Anti-CD137 for the Treatment of Surgically Resectable Pancreatic Adenocarcinoma
Brief Title: Comparing Neoadjuvant/Adjuvant GVAX vs a mKRASvax Given With Anti-PD-1 and Anti-CD137 for Surgically Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Agenus Inc. (Industry); Lustgarten Foundation (Other); Oncovir, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J24146; IRB00465956 (Other: Johns Hopkins Medicine Internal Review Board)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer
Keywords: Balstilimab; AGEN2373; KRAS peptide vaccine; peptide vaccine; Poly-ICLC; GVAX; Cyclophosphamide; Immunotherapy; Anti-PD-1 (anti-check point inhibitor); PD-L1 (check point inhibitor); Anti-CD137; Cancer vaccine; Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma (PDAC); Adenocarcinoma; Carcinoma; Pancreas; mKRASvax
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Carcinoma | interventions — balstilimab; Cyclophosphamide; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - AGEN2373/Balstilimab/Cyclophosphamide/GVAX (Experimental)
  Interventions: Drug: AGEN2373; Drug: Balstilimab; Drug: Cyclophosphamide; Drug: GVAX
- Arm 2 - AGEN2373/Balstilimab/mKRASvax (1.8mg total peptides +0.5mg each poly-ICLC) (Experimental)
  Interventions: Drug: AGEN2373 (RP2D); Drug: Balstilimab; Drug: mKRASvax

INTERVENTIONS:
Drug: AGEN2373 — 1. Up to 3 doses (1 mg/kg, 3 mg/kg, and 10 mg/kg) will be tested in Phase I to determine the dose to be used in Phase II. AGEN2373 will be administered as a 60 minute IV infusion (-5/+15 min) on Day 1 of each cycle for a total of 6 cycles of treatment. Cycle 1 (14 days) is prior to surgical resection, Cycle 2 (14 days) is after surgery and prior to standard of care chemotherapy, and Cycles 3-6 (21 days) are given after completion of chemotherapy.
  2. Drug: 1 mg/kg, 3 mg/kg, and 10 mg/kg IV
  Arms: Arm 1 - AGEN2373/Balstilimab/Cyclophosphamide/GVAX
Drug: Balstilimab — 1. 450 mg will be administered as a 30 minute IV Infusion (-5/+15 min) on day 1 of each cycle for a total of 6 cycles of treatment. Cycle 1 (14 days) is prior to surgical resection, Cycle 2 (14 days) is after surgery and prior to standard of care chemotherapy, and Cycles 3-6 (21 days) are given after completion of chemotherapy.
  2. Drug: 450 mg IV
  Other Names: AGEN2034, anti-PD-1 antibody
  Arms: Arm 1 - AGEN2373/Balstilimab/Cyclophosphamide/GVAX
Drug: Cyclophosphamide — 1. 200 mg/m2 will be administered as a 30 minute IV infusion (-5/+15 min) on day 1 of each cycle for a total of 6 cycles of treatment. Cycle 1 (14 days) is prior to surgical resection, Cycle 2 (14 days) is after surgery and prior to standard of care chemotherapy, and Cycles 3-6 (21 days) are given after completion of chemotherapy.
  2. Drug: 200 mg/m2 IV
  Other Names: Cy
  Arms: Arm 1 - AGEN2373/Balstilimab/Cyclophosphamide/GVAX
Drug: GVAX — 1. Vaccine (5 × 108 cells) will be administered on Day 2 of each cycle for a total of 6 cycles of treatment. Six intradermal injections will be given in the upper thighs and non-dominant arms. Cycle 1 (14 days) is prior to surgical resection, Cycle 2 (14 days) is after surgery and prior to standard of care chemotherapy, and Cycles 3-6 (21 days) are given after completion of chemotherapy.
  2. Drug: GVAX
  Other Names: PANC 10.05 pcDNA-1/GM-Neo vaccine and PANC 6.03 pcDNA-1/GM-Neo vaccine
  Arms: Arm 1 - AGEN2373/Balstilimab/Cyclophosphamide/GVAX
Drug: AGEN2373 (RP2D) — 1. Drug: Up to 3 doses (1 mg/kg, 3 mg/kg, and 10 mg/kg) will be administered as a 60 minute IV. Infusion (-5/+15 min) on Day 1 of each cycle for a total of 6 cycles of treatment. Cycle 1 (14 days) is prior to surgical resection, Cycle 2 (14 days) is after surgery and prior to standard of care chemotherapy, and Cycles 3-6 (21 days) are given after completion of chemotherapy.
  2. Drug: 1 mg/kg, 3 mg/kg, and 10 mg/kg IV
  Arms: Arm 2 - AGEN2373/Balstilimab/mKRASvax (1.8mg total peptides +0.5mg each poly-ICLC)
Drug: Balstilimab — 1. 450 mg will be administered as a 30 minute IV. Infusion (-5/+15 min) on day 1 of each cycle for a total of 6 cycles of treatment. Cycle 1 (14 days) is prior to surgical resection, Cycle 2 (14 days) is after surgery and prior to standard of care chemotherapy, and Cycles 3-6 (21 days) are given after completion of chemotherapy.
  2. Drug: 450 mg IV
  Other Names: AGEN2034, anti-PD-1 antibody
  Arms: Arm 2 - AGEN2373/Balstilimab/mKRASvax (1.8mg total peptides +0.5mg each poly-ICLC)
Drug: mKRASvax — 1. mKRASvax will be administered on Day 1 of each cycle and on Day 8 of Cycle 1 only. mKRASvax is given as 5 subcutaneous injections administered in the upper thighs and arms. Cycle 1 (14 days) is prior to surgical resection, Cycle 2 (14 days) is after surgery and prior to standard of care chemotherapy, and Cycles 3-6 (21 days) are given after completion of chemotherapy.
  2. 0.3 mg per peptide vaccine + 0.5mg Poly-ICLC
  Other Names: mutant KRAS peptide vaccine with Hiltonol® (Poly-ICLC)
  Arms: Arm 2 - AGEN2373/Balstilimab/mKRASvax (1.8mg total peptides +0.5mg each poly-ICLC)

SUMMARY:
The purpose of this study is to determine the optimal dose of AGEN2373 that is safe when given in combination with balstilimab and Pancreatic GVAX Whole Cell Vaccine and evaluate the safety and clinical activity of balstilimab and AGEN2373 in combination with GVAX (Arm 1) or mKRASvax (Arm 2) in surgically resectable pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Have a newly diagnosed, biopsy-proven adenocarcinoma of the pancreas.
* Tumor must be deemed resectable by the study team
* Patient's acceptance to have a tumor biopsy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests and procedures.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test.
* For both Women and Men, must use acceptable form of birth control while on study.

Exclusion Criteria:

* Received any anti-pancreatic cancer therapy (symptomatic therapies are allowed), or any prior anti-cancer immunotherapy.
* Diagnosed with another cancer whose natural history or treatment could interfere with safety or efficacy assessments on this study.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active autoimmune disease.
* Systemic steroid therapy (> 10mg daily prednisone equivalent) or immunosuppressive therapy within 14 days of first dose of study drug administration.
* Active infection requiring systemic therapy.
* Known history of human immunodeficiency virus (HIV).
* Active or chronic hepatitis B or hepatitis C.
* Known active tuberculosis.
* History of interstitial lung disease, non-infectious pneumonitis or uncontrolled lung diseases including pulmonary fibrosis, acute lung diseases, chronic obstructive pulmonary disease (COPD), asthma requiring medication, etc.
* Prior allogeneic stem cell transplantation or organ transplantation.
* Any major surgical procedure requiring general anesthesia ≤ 28 days before first dose of study drug.
* Received a live vaccine ≤ 28 days before first dose of study drug.
* History of severe hypersensitivity reaction to any monoclonal antibody
* Concurrent participation in another therapeutic clinical study
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities in Phase I participants | 1 month
  Phase I participants will be evaluated for dose limiting toxicities (DLTs) during the first 14 day cycle and 14 days post-operatively for the purpose of determining the recommended phase II dose of AGEN2373 when given concurrently with balstilimab and cancer vaccination.
Number of participants experiencing Grade 3 or Higher study drug-related toxicities | 2 years
  Number of participants experiencing study drug-related adverse events Grade 3 or higher as defined by CTCAE v5.0
Number of participants who form Intratumoral tertiary lymphoid structures (TLS) | 2 weeks
  Number of participants who form at least one tertiary lymphoid structure (TLS) following one cycle of study drugs. The presence of at least 50 CD20+ B cells and 50 CD3+ T cells in a ≥50 µM area of surgical tissue is considered "positive" for TLS.

SECONDARY OUTCOMES:
Pathologic overall response rate (pORR) | evaluated at time of surgery, approximately 2 weeks from first dose of study drug
  Number of participants who have a pathologic response to the first dose of study drug as determined using surgically resected tissue and the College of American Pathologists (CAP) scoring system. A pathologic response is defined as CAP grade of 0-2. Possible CAP grades include grade 0: Complete Response/ No viable residual tumor; grade 1: Marked Response/ minimal residual cancer with single cells or small groups of cancer cells; grade 2: Moderate Response/ residual cancer outgrown by fibrosis; and grade 3: Poor or No response/ extensive residual cancer.
CD3+CD8+CD137+ T cell density in Tumor Tissue | evaluated at time of surgery, approximately 2 weeks from first dose of study drug
  Number of CD3+CD8+CD137+ T cells found in resected surgical tissue by Immunohistochemistry (IHC).
Change in peripheral interferon-gamma (IFNγ) producing mutant KRAS-specific T cells | 13 weeks
  Percent change in the number of IFNγ producing T cells at Cycle 2 Day 14 when compared with baseline. Number of IFNγ T cells will be assessed by ELISPOT.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Christenson, MD, Principal Investigator — SKCCC • Johns Hopkins Medical Institution
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No